CLINICAL TRIAL: NCT07003750
Title: Surgical Wound Infection Prevention Bundle in Patients Undergoing Coronary Bypass Graft Surgery Sohag Experience
Brief Title: Surgical Wound Infection Prevention Bundle in Patients Undergoing Coronary Bypass Graft Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ragab Mostafa, cardiothoracic surgery resident, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: soh-Med--25-4-05MS
Record Dates: First submitted 2025-05-08; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Infection Due to Coronary Artery Bypass Graft (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): * Preoperative:
    1. Nightly CHG baths
    2. Mupirocin nasal ointment twice daily for 2 to 5 days prior to surgery
    3. Hair removal with clippers
  * Intraoperative:
    1. Skin antisepsis with CHG solution
    2. Standardized IV antibiotic doses at the following time points :within 5 to 60 minutes of the initial surgical incision, with initiation of cardiopulmonary bypass ,and every 3 hours intraoperatively for the duration of the case.
  * Postoperative :
    1. The occlusive sternal dressing applied at time of chest closure and removed 48 hours postoperatively then daily dressing thereafter.
    2. Daily postoperative linen change and minimize sternotomy exposure to home blankets
  Interventions: Other: Surgical wound infection prevention bundle
- group 2 (No Intervention): * Preoperative:
    1. Preoperative water and soap bath
    2. Hair removal with razor
  * Intraoperative:
    1. Skin antisepsis with betadine solution
    2. One dose of antibiotic just before skin incision
  * Postoperative:
    1. The occlusive sternal dressing removed 72 hours postoperatively then daily dressing
    2. No specific concerns about linens change and home blankets exposure

INTERVENTIONS:
Other: Surgical wound infection prevention bundle — utilization of locally customized surgical wound infection bundle to prevent and or control of infection in patients undergoing CABG surgery
  Arms: group 1

SUMMARY:
estimate the utilization of locally customized surgical wound infection bundle to prevent and or control of infection in patients undergoing CABG surgery in Sohag

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease ,diebetes mellitus,hypertension,

Exclusion Criteria:

* patients who have cancer , immunocompromised patients, cardiac surgeries other than CABG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
surgical site wound infection | From enrollment to 6 months after surgery
  Early complications including superficial and deep surgical site infection. Late complications including DSWI, systemic and chronic sinus

IPD SHARING:
Plan to Share IPD: No